CLINICAL TRIAL: NCT05684809
Title: Efficacy of Cervical Mobilization With Post Isometric Relaxation in Managing Mechanical Neck Pain Associated With Myofascial Trigger Points: a Randomized Comparative Study
Brief Title: Efficacy of Mobilization With Post- Isometric Relaxation in Neck Pain Associated With Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Najran University (Other)
Responsible Party: Principal Investigator, Hashim Ahmed, Assistant Professor, Najran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 444-42-20993-DS
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Mechanical Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): in addition to Conventional treatment, PIR and cervical mobilization were given
  Interventions: Other: Post Isometric relaxation Technique (PIR); Other: Cervical Mobilization (CM); Other: conventional treatment
- Group B (Active Comparator): in addition to Conventional treatment, PIR were given
  Interventions: Other: Post Isometric relaxation Technique (PIR); Other: conventional treatment

INTERVENTIONS:
Other: Post Isometric relaxation Technique (PIR) — In PIR intervention, the patients were requested to lie down in a supine position and their neck was in a lateral flexion to the opposite side so that the target upper Trapezius muscle fibers would be in a lengthened position. The therapist performed a moderate isometric contraction (approximately 75% of maximal) of upper Trapezius muscles, held it for 5 seconds, then relaxed for 3 seconds before moving the cervical spine into the new barrier. In each session, this technique was repeated for four times, on alternate days for three weeks.
Other: Cervical Mobilization (CM) — Cervical Mobilization was delivered in prone lying with their foreheads resting comfortably on his hands, and the chin was tucked in.The treatment session was done on alternate days (3 days a week) for 3 weeks, hence the total number of sessions were 9.
  Arms: Group A
Other: conventional treatment — Hot Pack was given for twenty minutes, slow sustained stretching exercises ( 20 second hold, 10-second relaxation) were given, and isometric exercise of the neck((10 repetitions of two sets with 10 seconds hold) alternate days for three weeks.

SUMMARY:
purpose of the study: to determine the effectiveness of cervical mobilization with PIR in reducing pain and improving neck ROM and function in people with mechanical neck pain associated with MTrPs

DETAILED DESCRIPTION:
This study will be based on a randomized controlled design which will be comparative in nature. Participants will be recruited using the convenience sampling method and will be randomly divided into two groups A and B respectively. Thirty participants of mechanical neck pain associated with upper Trapezius trigger point pain will be recruited from the Physiotherapy department, at the Najran University, Saudi Arabia. Study objectives and procedure will be properly explained and written informed consent will be obtained at the beginning of the study. All the participants will be randomly assigned into two equal groups A and B.

Group A will be receiving the hot pack, active Stretching, isometric exercise intervention, and PIR technique while group B will receive the hot pack, active Stretching, isometric exercise intervention, and cervical Mobilization.

ELIGIBILITY:
Inclusion Criteria:

* age 20-40 years,
* having mechanical neck pain located in the neck or scapular regions along with 1-2 MTrPs which,
* on palpation replicated their chief complaints in the upper Trapezius muscle (unilateral).

Exclusion Criteria:

* known cases of fibromyalgia syndrome,
* cervical radiculopathy or myelopathy,
* history of cervical spine surgery,
* congenital or acquired postural deformity, presence of MTrPs in bilateral upper Trapezius muscles,
* patients who received any treatment for their pain one month prior to the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 3 Weeks
  The pain intensity was assessed Using a numeric pain rating scale (NPRS), Its a 11 point scale, where zero indicates no pain and 10 indicates severe pain
Neck Disability Index | 3 Weeks
  The Neck Disability was assessed using a neck disability index (NDI) questionnaire, the minimum value 0- and the maximum value is 50
Range of Motion | 3 Weeks
  The Neck Side Flexion range of motion was assessed using cervical range of motion(CROM) device
Pain Pressure Threshold | 3 Weeks
  The Pain Pressure Threshold (PPT) was assessed using an algometer algometer

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Ahmed, PhD, Principal Investigator — Najran University
Locations (1):
- Hashim Ahmed, Najrān, Najran Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No